CLINICAL TRIAL: NCT03951909
Title: Effect of Physiotherapy and Psychological Group Treatment on Physical and Mental Health Among Refugees From Syria With Pain Disorders or Post-traumatic Symptoms
Brief Title: Physiotherapy and Psychological Among Refugees From Syria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Bergen (Other)
Collaborators: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/603
Record Dates: First submitted 2019-02-15; First posted 2019-05-16 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pain; Mental Health Impairment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants identified with pain disorders or post-traumatic mental health symptoms according to previously defined objective selection criteria will be invited to the appropriate treatment group conducted by physiotherapists (for those with pain disorders) or health professionals trained in TRT techniques (for those with post-traumatic symptoms). Participants presenting both pain and post-traumatic symptoms will be invited to the intervention treatment for the symptom in which they score highest.
  For each group a waiting-list group receiving the same treatment some weeks later was the control group.
Masking Description: Neither the participant or th researcher knew the intervention assignment before enrollment, but there were no masking afterwards (when they had been assigned to either physiotherapy or TRT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): Either Physiotherapy activity and awareness intervention (PAAI) or Teaching recovery techniques (TRT)
  Interventions: Behavioral: Physiotherapy activity and awareness intervention: PAAI; Behavioral: Psychological intervention: Teaching recovery techniques (TRT)
- Waiting list (Experimental): The same interventions as above will be hold for waiting lists participants, but after 6 to 8 weeks
  Interventions: Behavioral: Physiotherapy activity and awareness intervention: PAAI; Behavioral: Psychological intervention: Teaching recovery techniques (TRT)

INTERVENTIONS:
Behavioral: Physiotherapy activity and awareness intervention: PAAI — 10 to 12 persons will be invited to each group. The intervention will consist on 8 weekly sessions including the same key elements each time: introduction with a mindfulness exercise and a ball game, several movements while sitting on a chair, standing proprioceptive exercises with wooden sticks and exercises to raise awareness of muscle tensions in the body, active movements stimulating the balance, coordination and breathing and finally relaxation and a short closing round.
Behavioral: Psychological intervention: Teaching recovery techniques (TRT) — TRT is composed of five two-hour group teaching sessions with up to 15 participants. The first two sessions deal with intrusive thoughts and feelings: problems such as bad memories, nightmares, and flashbacks. The third session deals with arousal, coming to the surface as difficulties in relaxing, concentrating and sleeping. The fourth and fifth sessions deal with avoidance: ones fears, and difficulties in facing up to reminders of the war and violence.

SUMMARY:
The war in Syria began in 2011 and refugees from this country have faced stressors including security risks, lack of access and availability of basic services and resources as well as family, community, and socio political tensions. Exposure to stressful events or situations, either short or long lasting, of exceptionally threatening or catastrophic nature is likely to cause pervasive distress in almost anyone, which might disturb daily life function, integration in society and ability to function in work and society, although this stress does not necessarily need to become an established medical diagnose. For a long time now, somatic and mental health systems have been overburdened and inaccessible both in Syria and in transit countries, and there is little available evidence of the effect of interventions targeting common health problems among refugees once established in their host countries.

In this project, the University of Bergen, in close collaboration with the Centre for Migration Health (Bergen municipality) and the Centre for Crisis Psychology, have developed two treatment interventions that are both theoretically sound and practically scalable if shown to be effective.

Among resettled asylum seekers and refugees, the primary aim of the project is to separately study in a quantitative way the effect on both physical and mental health of two different interventions: Physiotherapy activity and awareness intervention for participants with pain disorders and Teaching recovery techniques for participants with post-traumatic symptoms In addition, in a qualitative mode, our secondary aim is to analyse the processes by which the interventions help/do not help the patients to improve their health. Last, as the third aim of the study, cost effectiveness analyses will be conducted.

DETAILED DESCRIPTION:
Introduction Syria is now the 11th country of origin for immigrants in Norway. During the last two years, the numbers of asylum seekers from Syria with permanent refugee status have rapidly grown from 9700 in 2016 to a total of 20800 registered by the 1st of January 2017. Given that more than 1 million Syrians applied for asylum in Europe between April and December 2017, the numbers are probably going to continue growing also in Norway in the months to come.

Impact of stress on health The war in Syria began in 2011 and refugees from this country have faced stressors including security risks, lack of access and availability of basic services and resources as well as family, community, and socio political tensions. Exposure to stressful events or situations, either short or long lasting, of exceptionally threatening or catastrophic nature is likely to cause pervasive distress in almost anyone, which might disturb daily life function, integration in society and ability to function in work and society, although this stress does not necessarily need to become an established medical diagnose. For a long time now, somatic and mental health systems have been overburdened and inaccessible both in Syria and in transit countries. Although our knowledge of the health needs of refugees is still incomplete, several studies suggest a high degree of chronic pain disorders and mental health symptoms as a result of the previous factors.

Arthrosis, arthritis and other forms for chronic pain are especially disabling among the chronic non-communicable diseases and have previously been described to be related to mental health problems. Though there is a lack of data regarding these conditions, some available studies point to a relatively high prevalence among refugees from Syria. Just to point out some examples: Among young Syrian refugees attending an emergency department in Austria between 2011 and 2014, 12% presented chronic musculoskeletal problems and 9% suffered from chronic headaches. A cross-sectional survey of 1550 refugees conducted outside of camps in Jordan found a prevalence of 7% of arthritis. In the previously referred paper on elderly Syrians, 47% reported difficulty walking.

Regarding mental problems, 61% of older refugees from Syria living in Lebanon in 2011-2013 reported feeling anxious, and significant proportions reported feelings of depression, loneliness, and believing they were a burden to their families. In another study, 44% of 310 Syrian forced migrants in Lebanon in 2011 suffered from depression. In 2014, 54% of Syrians accessing International Medical Corps facilities in Syria and neighbouring countries suffered severe emotional disorders, including depression and anxiety.

Once resettled in Norway, the municipalities have the responsibility to offer adequate health care services to refugees in need of health care. However, lack of evidence regarding the best treatment together with limited resources may compromise the offer given to refugees. Group treatment can be a strategy to maximize the effect of the treatment given the resources typically available at the municipalities for this group of patients, as well as a mean to increase social interaction and well-being among participants.

Evidence on group-based physiotherapy on chronic pain among refugees is scarce. A study using basic body awareness therapy versus mixed physical activity for refugees with post traumatic stress disease (PSTD) is on-going in Denmark, but the authors chose to give personal treatment as opposed to group treatment due to a higher level of disease among their included participants. Norwegian group psychomotor physiotherapy and general physiotherapy exercises, on the other side, are well known and used in the Nordic countries. By using the knowledge of the body and reactions after trauma, the physiotherapist can recognize and normalize the participants emotions and movement patterns, capturing and preserving the individual needs within the group, at the same time as having an overview of the group and the social interactions within it.

Teaching recovery techniques (TRT) is a group-based mental health intervention developed by the Children and war foundation to use on subjects exposed to war or nature catastrophes previously used in the Centre for migration and health at the municipality of Bergen. This treatment addresses the three main trauma symptoms: intrusion, arousal and avoidance. Several studies on the effect of TRT have been carried out with children surviving catastrophes and adolescent asylum seekers in Europe, all showing significant reductions in established mental health disorders (PTSD). Among adolescents in Palestine, TRT has recently been shown to significantly reduce posttraumatic stress symptoms and was evaluated as a cost-effective intervention. However, as far as theinvestigators know the effect on TRT has not previously been studied in an adult population with post-traumatic symptoms.

Our hypotheses for the development of the interventions are the following: Among asylum seekers and refugees resettled in Norway

* Pain disorders and post-traumatic symptoms often coexist and are related to each other
* Group physiotherapy treatment reduces pain levels
* Group physiotherapy treatment improves mental health
* Self-help groups using TRT improve mental health
* Self-help groups using TRT reduce pain levels
* Social and contextual factors and previous migration experiences are related to the effect of treatment

Aims of the study

Among resettled asylum seekers and refugees, the primary aim is to separately study in a quantitative way the effect on both physical and mental health of two different interventions:

1. Physiotherapy activity and awareness intervention (PAAI) for participants with pain disorders
2. TRT for participants with post-traumatic symptoms In addition, in a qualitative mode, our secondary aim is to analyse the processes by which the interventions help/do not help the patients to improve their health. Last, as the third aim of the study, cost effectiveness analyses will be conducted.

Interventions Two different interventions have been developed in close collaboration with all collaborating parts and based in both theory and experience.

1. Physiotherapy activity and awareness intervention: PAAI The physiotherapy treatment will be held in groups based on principles from the Norwegian psychomotor physiotherapy and general physiotherapy exercises.
2. Psychological intervention: Teaching recovery techniques (TRT) The mental health self-help groups are based on the manual TRT developed by Children and war foundation based on Trauma focused cognitive behavioural Therapy. Each group will be conducted by two members of the team. An effort has been done to certify collaborating interpreters and the investigators will try to use the same interpreters for a given group. TRT is designed to teach children in a step-by-step practical way to develop some skills and techniques helpful in coping with the psychological effects of war and violence.

Study design Our study is designed as a randomised trial comparing the intervention with a control arm. The control arm will be offered the same intervention after a time lag enabling comparison (waiting-list-control trial). This design enables assessment of the intervention and has practical advantages in implementation. The same design will be used for both the PAAI and the TRT intervention. Participants with predominantly pain symptoms will be invited to the PAAI intervention and participants with predominantly post-traumatic symptoms will be invited to the TRT intervention. Participants scoring high on both symptoms will be offered the intervention for which they score highest in the respective symptoms scales. Once assessed for eligibility and given informed consent as explained above, randomisation of each participant to the appropriate trial will be conducted (individualised 1:1 randomisation into groups). Participants will be randomised to the immediate intervention group (IIG) or to a waiting list control group (WLG). The WLG will receive usual care during the first 7/8 weeks, depending on the intervention, at which point they will cross over to the intervention arm and receive the intervention for 7/8 weeks. Both groups will be reassessed 12 weeks after the intervention.

In addition to the assessment of the effect of the intervention through quantitative methods as described under, an embedded qualitative process evaluation will be organised to learn how the interventions are perceived by the target group and the therapists, and receive input to make the necessary adjustments.

ELIGIBILITY:
Inclusion Criteria:

• Patients who answer yes to the question "Have you experienced any of these or some other terrifying event(s)?" and score over 24 in the revised Impact of Events Scale (R-IES) will be invited to the TRT-intervention.

Exclusion Criteria:

* Patients who report health conditions requiring close medical follow up
* Patients who score in the mental health questions as having a serious mental illness (37 + in the revised Impact of Events Scale or 25 or more in the GHQ-12)
* Patients with a living situation that impedes following up (including no current address close to Bergen).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in body pain index using Body Pain Inventory | At recruitment, right before and after the intervention and 12 weeks afterwards
  Pain intensity measures through four questions: worst pain, least pain, average pain, pain right now). Each question can answers with 1 to 10 points and will be measured separately
Change in Impact of Events Scale | At recruitment, right before and after the intervention and 12 weeks afterwards
  Scores in the Impact of Events-Revised scale. The revised version of the Impact of Event Scale has 22 questions and a scoring range of 0 to 88. Low scores are considered as better outcomes. Scores of 24 or more are of clinical concern and 33 and above is the cutoff for a probable diagnoses of post traumatic stress disorder(PTSD)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No
Sensitive information. Not allowed to share by the Ethical committee

REFERENCES:
- [Derived] Hasha W, Igland J, Fadnes LT, Kumar BN, Heltne UM, Diaz E. Effect of a self-help group intervention using Teaching Recovery Techniques to improve mental health among Syrian refugees in Norway: a randomized controlled trial. Int J Ment Health Syst. 2022 Sep 6;16(1):47. doi: 10.1186/s13033-022-00557-4. PMID 36068576
- [Derived] Hasha W, Fadnes LT, Igland J, Vardal R, Giusti LM, Stromme EM, Haj-Younes J, Heltne U, Kumar BN, Diaz E. Two interventions to treat pain disorders and post-traumatic symptoms among Syrian refugees: protocol for a randomized controlled trial. Trials. 2019 Dec 27;20(1):784. doi: 10.1186/s13063-019-3919-x. PMID 31881990
- See also: Description of the CHART study, of which this project is the RCT part — https://www.uib.no/en/generalpractice/chart